CLINICAL TRIAL: NCT04608149
Title: Carpediem(TM) Post Market Surveillance Study
Brief Title: Prospective, Multi-center, Single-arm, Observational Study. US FDA 522 Pediatric Post Market Surveillance Study.
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20039
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Kidney Injury; Fluid Overload
Keywords: Carpediem(tm); continuous renal replacment therapy; CRRT; acute kidney injury; pediatric; fluid overload; hemodialysis; hemofiltration; post market surveillance; registry
MeSH Terms: conditions — Acute Kidney Injury; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects treated with Carpediem system: All patients who receive CRRT with the Carpediem™ system, as prescribed by the investigator, will be offered participation in the post market surveillance study after obtaining parental consent.
  Interventions: Device: Carpediem System

INTERVENTIONS:
Device: Carpediem System — Continuous renal replacement therapy

SUMMARY:
The post market surveillance study will employ a prospective, multi-center, single-arm, observational design to capture data on children who undergo CRRT using the Carpediem™ system. Participating clinicians will manage subjects in accordance to their local standard of care practices and decisions on initiating, modifying or discontinuing CRRT are up to the local investigative team's prescription.

A minimum of 10 centers in the United States, that have been trained on the use of the Carpediem™ system, will be invited to participate in the study. After obtaining institutional review board approval and written informed consent from a parent or legally authorized representative (LAR), data from all subjects treated with the Carpediem™ system will be included in the study. A minimum of 35 subjects will be enrolled and sites may be asked to screen and enroll patients for the study for up to 36 months.

Status of subjects discharged from hospital will be collected at 30- and-90 days following hospital discharge by phone interviews in accordance to local standard of care practices, review of in-hospital records or in-clinic visit, as available.

DETAILED DESCRIPTION:
The post market surveillance study is designed to capture data in the real-world clinical setting on the use of the Carpediem™ system and will evaluate the safety and performance in children requiring CRRT in the US. Data on survival and the effectiveness of the Carpediem™ system on renal function recovery will be evaluated. A comprehensive evaluation of subjects being treated with Carpediem™ will include, but is not limited to, acuity at hospital/ICU admission and prior to CRRT initiation, Carpediem™ treatment parameters, laboratory data, and requirement for mechanical ventilation and/or inotropic support. Subject status and requirement for renal replacement therapy post hospital discharge will be evaluated at 30- and 90-days.

ELIGIBILITY:
Inclusion Criteria:

* Parent or LAR has signed information consent
* Subject weighs between 2.5-10 kg (or 5.5-22 lbs)
* Subject is receiving medical care in an intensive care unit
* Parental or LAR consent to receive full supportive care through aggressive management utilizing all available therapies for a minimum of 96 hours
* Subject has a clinical diagnosis of acute kidney injury per Kidney Disease Improving Global Outcomes (KDIGO) criteria or fluid overload requiring CRRT

Exclusion Criteria:

* Subject is not expected to survive 72 hours due to an irreversible medical condition, in the opinion of the investigator
* Subject has irreversible brain damage, in the opinion of the investigator
* Subject is intolerant to anticoagulation, as documented in the medical record
* Subject has a Do Not Attempt Resuscitate (DNAR), Allow Natural Death (AND), withdrawal of care or similar order, or anticipated change in status, in the opinion of the investigator, within the next 7 days
* Subject has pre-existing end-stage renal disease or pre-existing, advanced chronic kidney disease, defined as an estimated Glomerular Filtration Rate (eGRF) < 30 ml/min/1.73m2
* Subject is currently or has chronically been treated with a circulatory support device (i.e., left ventricular assist device (LVAD)) other than ECMO
* Subject has had prior CRRT treatments using the Carpediem™ system
* Subject is enrolled in clinical trials or being treated with other investigational therapeutic devices or products for acute kidney injury or fluid overload
* Subject has any other medical condition that may confound the study objectives, in the opinion of the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have acute kidney injury or fluid overload requiring hemodialysis or hemofiltration who weigh between 2.5 and 10 kilograms (5.5 to 22 pounds).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Survival at CRRT Discontinuation | from the start of CRRT to the date of death or CRRT discontinuation, assessed up to 100 weeks
  Evaluation subject survival at CRRT discontinuation
Survival at intensive care unit (ICU) discharge | from the start of CRRT to the date of death or ICU dhscharge, assessed up to 100 weeks
  Evaluation subject survival at ICU discharge

SECONDARY OUTCOMES:
Survival through 90 days post hospital discharge | hospital discharge through 90 days post discharge
  Quantify survival at hospital discharge, and 30- and 90-days post hospital discharge
Hospital and ICU length of stay | through discharge, assessed up to 100 weeks
  Evaluation hospital and ICU length of stay
Renal function recovery at discharge and 30- and 90- days post hospital discharge | Hospital discharge through 90 days post discharge
  Assess renal function recovery at hospital discharge and 30- and 90- days post hospital discharge
Overall survival | through study completion, an average of 3 years
  Characterize overall survival based on variables including, but not limited to; demographic data, laboratory values, patient acuity prior to CRRT initiation and CRRT treatment parameters
Time to CRRT discontinuation | from the start of CRRT to the date of death or CRRT discontinuation, assessed up to 100 weeks
  Assess time to CRRT discontinuation
Carpediem system-related adverse events | through study completion, an average of 3 years
  Quantify the rate of Carpediem system-related adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Iowa Healthcare, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Golisano Children's Hospital, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No